CLINICAL TRIAL: NCT01680224
Title: Effectiveness Trial of a Dissonance-Based Obesity Prevention Program
Acronym: Project Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HD071900
Record Dates: First submitted 2012-08-29; First posted 2012-09-07 (Estimated); Last update posted 2018-09-21 (Actual); Status verified 2018-09

CONDITIONS: Obesity; Weight Gain; Eating Disorders
Keywords: Obesity; Weight Gain; Dissonance; College,University Students; Eating Disorders; Obesity Prevention; Selective Prevention; Effectiveness
MeSH Terms: conditions — Obesity; Weight Gain; Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Healthy Weight (Active Comparator): The main goal of the Healthy Weight intervention is to make small, sustainable changes to input and output on a weekly basis to achieve a balance between caloric intake and output. All sessions begin with a brief review of what was covered in the previous session, presentation of educational handouts, careful review of previous behavior change goals, and the development of healthy behavior change plans for the next session. Home exercises for all sessions consist of following individualized diet and exercise goals, and keeping a food and exercise log to determine areas for future healthy changes.
  Interventions: Behavioral: Healthy Weight
- Project Health (Experimental): Project Health adds dissonance-inducing activities, discussions, and homework activities to the Healthy Weight basic intervention. Each session begins with a verbal commitment to participate (to underscore the voluntary nature of participation), includes discussions of completed home practice assignments and in-session writing/sharing exercises (to create accountability), and concludes with home exercises (to increase level of effort). Completed home assignments are videotaped in subsequent sessions to increase accountability.
  Interventions: Behavioral: Project Health
- Control (Placebo Comparator): Some participants will be randomized to control condition whereby they will be given an psychoeducational video ("Weight of the World")to view.
  Interventions: Behavioral: Placebo Control

INTERVENTIONS:
Behavioral: Healthy Weight
  Arms: Healthy Weight
Behavioral: Project Health
  Arms: Project Health
Behavioral: Placebo Control — Participants will view a video on overweight and obesity
  Arms: Control

SUMMARY:
Obesity is a major US public health problem. Few obesity prevention programs have reduced risk for weight gain over follow-up and those that have are very intensive, making dissemination difficult and costly. A brief 3-hr selective prevention program (Healthy Weight) targeting young adults with body dissatisfaction involving participant-driven healthy dietary and physical activity lifestyle changes significantly reduced increases in body mass index (BMI) and obesity onset relative to alternative interventions and assessment-only controls through 3-yr follow-up, though effects were small in magnitude. To enhance efficacy, the investigators added dissonance-inducing activities regarding unhealthy dietary and activity practices, drawing from a highly efficacious dissonance-based eating disorder prevention program. A pilot trial found that this new Project Health intervention significantly reduced increases in BMI relative to both the Healthy Weight intervention and an educational brochure condition from pre to post. The investigators propose to conduct a rigorous multisite effectiveness trial that will test whether adding the dissonance-induction elements to the originally Healthy Weight intervention improves weight gain prevention effects. 360 college students at risk for future weight by virtue of their age and weight concerns will be randomized one of three conditions: (1) a refined 6-hr group-based dissonance-based Project Health, (2) a 6-hr group-based Healthy Weight intervention, or (3) a psychoeducational video ("Weight of the World") condition. Participants will complete assessments of % body fat, mediators (including objectively measured physical activity), moderators, and other outcomes at pre, post, and 6, 12, and 24 month follow-ups.

DETAILED DESCRIPTION:
Aim 1 will test the hypothesis that Project Health significantly reduces increases in % body fat relative to the Healthy Weight intervention and video control condition during a 2-yr follow-up; secondary outcomes are BMI, depressive symptoms and eating disorder symptoms. The investigators will also compare Healthy Weight to video controls.

Aim 2 will test the hypothesis that Project Health participants will experience increased cognitive dissonance (an uncomfortable psychological state) regarding eating unhealthy foods and engaging in sedentary behaviors, and that changes in dissonance mediate the program's weight gain prevention effects. The investigators will also test whether reduced calorie intake and increased physical activity mediate the effects of Project Health on change in % body fat.

Aim 3 will test the hypothesis that intervention effects are amplified for participants with elevated body dissatisfaction (which should increase motivation change) and preference for consistency (which should maximize dissonance induction) and mitigated for participants who report emotional eating and substance use (because these factors increase risk for overeating).

ELIGIBILITY:
Inclusion Criteria:

* University student
* Presents with self-reported "weight concerns"

Exclusion Criteria:

* Diagnosis of Eating Disorder
* Obese
* Underweight
* Non-english speaking

Ages: 17 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 364 (Actual)
Dates: Start 2012-09-01 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Body Fat Percentage | Changes in body fat from baseline to 2-year follow up
  We will use air displacement plethysmography (ADP) via the Bod Pod S/T to assess % body fat. Two measures will be averaged. Body density, calculated as body mass divided by estimated body volume, is used to calculate age- and gender-adjusted body fat percentile scores, based on normative reference data (McCarthy et al., 2006). A pilot validity study (N = 30) revealed that direct DEXA measures of % body fat correlates much more strongly with ADP estimates of body fat (r = .88) than with BMI (r = .23). Change in age- and gender-adjusted body fat percentile over the 2-year follow-up will be the primary outcome. This assessment takes 3-5 minutes to complete.

SECONDARY OUTCOMES:
Eating Pathology | Baseline and post intervention (6 weeks); 6/12/24 month follow-up
  The Eating Disorder Diagnostic Interview, a brief semi-structured interview, will assess eating disorder symptoms. It provides diagnoses for anorexia nervosa, bulimia nervosa, and binge eating disorder, which will allow us to exclude participants with these disorders. It also provides a continuous measure of overall eating disorder symptoms.
Negative Affect | Baseline and post intervention (6 weeks); 6/12/24 month follow-ups
  The 20-item Negative Affect subscale of the Positive and Negative Affect Schedule (PANAS: Watson et al., 1988) measures general negative affectivity and depressive symptoms. Using a Likert rating system, participants choose their degree of endorsement of negative affectivity items such as "disgusted with self" and "lonely" (response options: 1 = not at all; 5 = extremely).
Food Craving/Liking | Baseline, 6 weeks (post intervention), 6/12/24 month follow ups
  The 28-item Food Craving Inventory (FCI; White et al., 2002) assesses subjective cravings for individual foods (pasta, ice cream), asking: "Over the past month, how often have you experienced a craving for the food?"

OTHER OUTCOMES:
Weighing Habits | Baseline and post intervention (6 weeks); 6/12/24 mo follow-ups
  Participants will be asked how often they weighed themselves "in the past two weeks" at each assessment.
Physical Activity | Baseline and post-intervention (6 weeks); 6/12/24 month follow-ups
  Accelerometers will give objective measures of physical activity from each participant at each wave assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Stice, PhD, Principal Investigator — Oregon Research Institute; Paul Rohde, PhD, Study Director — Oregon Research Institute; Heather Shaw, PhD, Study Director — Oregon Research Institute; Kyle Burger, PhD, Study Director — Oregon Research Institute; Nathan Marti, PhD, Study Director — Oregon Research Institute
Locations (4):
- United States (4):
  - Oregon State University, Corvallis, Oregon
  - University of Oregon, Eugene, Oregon
  - Oregon Research Institute, Eugene, Oregon
  - University of Texas, Austin, Austin, Texas

REFERENCES:
- [Background] Anderson DA, Shapiro JR, Lundgren JD. The freshman year of college as a critical period for weight gain: an initial evaluation. Eat Behav. 2003 Nov;4(4):363-7. doi: 10.1016/S1471-0153(03)00030-8. PMID 15000962
- [Background] Becker CB, Stice E, Shaw H, Woda S. Use of empirically supported interventions for psychopathology: can the participatory approach move us beyond the research-to-practice gap? Behav Res Ther. 2009 Apr;47(4):265-74. doi: 10.1016/j.brat.2009.02.007. Epub 2009 Feb 21. PMID 19281965
- [Background] van den Berg P, Neumark-Sztainer D. Fat 'n happy 5 years later: is it bad for overweight girls to like their bodies? J Adolesc Health. 2007 Oct;41(4):415-7. doi: 10.1016/j.jadohealth.2007.06.001. PMID 17875468
- [Background] Blair AJ, Lewis VJ, Booth DA. Does emotional eating interfere with success in attempts at weight control? Appetite. 1990 Oct;15(2):151-7. doi: 10.1016/0195-6663(90)90047-c. PMID 2268140
- [Background] Block G, Subar AF. Estimates of nutrient intake from a food frequency questionnaire: the 1987 National Health Interview Survey. J Am Diet Assoc. 1992 Aug;92(8):969-77. PMID 1640041
- [Background] Bohon C, Stice E, Spoor S. Female emotional eaters show abnormalities in consummatory and anticipatory food reward: a functional magnetic resonance imaging study. Int J Eat Disord. 2009 Apr;42(3):210-21. doi: 10.1002/eat.20615. PMID 19040270
- [Background] Block G, Hartman AM, Naughton D. A reduced dietary questionnaire: development and validation. Epidemiology. 1990 Jan;1(1):58-64. doi: 10.1097/00001648-199001000-00013. PMID 2081241
- [Background] Boomsma. (2000). Reporting analyses of covariance structures. Structural Equation Modeling, 7, 461-483.
- [Background] Boutelle KN, Hannan P, Fulkerson JA, Crow SJ, Stice E. Obesity as a prospective predictor of depression in adolescent females. Health Psychol. 2010 May;29(3):293-8. doi: 10.1037/a0018645. PMID 20496983
- [Background] Burton E, Stice E. Evaluation of a healthy-weight treatment program for bulimia nervosa: a preliminary randomized trial. Behav Res Ther. 2006 Dec;44(12):1727-38. doi: 10.1016/j.brat.2005.12.008. Epub 2006 Feb 3. PMID 16458252
- [Background] Butler SM, Black DR, Blue CL, Gretebeck RJ. Change in diet, physical activity, and body weight in female college freshman. Am J Health Behav. 2004 Jan-Feb;28(1):24-32. doi: 10.5993/ajhb.28.1.3. PMID 14977156
- [Background] Chambers WJ, Puig-Antich J, Tabrizi MA, Davies M. Psychotic symptoms in prepubertal major depressive disorder. Arch Gen Psychiatry. 1982 Aug;39(8):921-7. doi: 10.1001/archpsyc.1982.04290080037006. PMID 7103681
- [Background] Cialdini, R. B., Trost, M. R., & Newsom, J. T. (1995). Preference for consistency: The development of a valid measure and the discovery of surprising behavioral implications. J Pers Soc Psychol, 69, 318-328.
- [Background] Coleman KJ, Tiller CL, Sanchez J, Heath EM, Sy O, Milliken G, Dzewaltowski DA. Prevention of the epidemic increase in child risk of overweight in low-income schools: the El Paso coordinated approach to child health. Arch Pediatr Adolesc Med. 2005 Mar;159(3):217-24. doi: 10.1001/archpedi.159.3.217. PMID 15753263
- [Background] Colley RC, Tremblay MS. Moderate and vigorous physical activity intensity cut-points for the Actical accelerometer. J Sports Sci. 2011 May;29(8):783-9. doi: 10.1080/02640414.2011.557744. PMID 21424979
- [Background] Cummins S, Macintyre S. Food environments and obesity--neighbourhood or nation? Int J Epidemiol. 2006 Feb;35(1):100-4. doi: 10.1093/ije/dyi276. Epub 2005 Dec 7. No abstract available. PMID 16338945
- [Background] Dietz WH, Robinson TN. Use of the body mass index (BMI) as a measure of overweight in children and adolescents. J Pediatr. 1998 Feb;132(2):191-3. doi: 10.1016/s0022-3476(98)70426-3. No abstract available. PMID 9506622
- [Background] Eisenberg, N., Cialdini, R. B., McCreath, H., Shell, R. (1989). Consistency-based compliance in children: when and why do consistency procedures have immediate effects? International Journal of Behavioral Development, 12, 351-367.
- [Background] Ello-Martin, J. A., Roe, L., & Rolls, B. (2004). A diet reduced in energy density results in greater weight loss than a diet reduced in fat. Obes Res, 12, A23-A23.
- [Background] Esliger DW, Probert A, Connor Gorber S, Bryan S, Laviolette M, Tremblay MS. Validity of the Actical accelerometer step-count function. Med Sci Sports Exerc. 2007 Jul;39(7):1200-4. doi: 10.1249/mss.0b013e3804ec4e9. PMID 17596790
- [Background] Esliger DW, Tremblay MS. Technical reliability assessment of three accelerometer models in a mechanical setup. Med Sci Sports Exerc. 2006 Dec;38(12):2173-81. doi: 10.1249/01.mss.0000239394.55461.08. PMID 17146326
- [Background] Everitt, B., & Pickles, A. (2004). Statistical aspects of the design and analysis of clinical trials. London: Imperial College Press.
- [Background] Festinger, L. (1957). A theory of cognitive dissonance. Stanford University Press.
- [Background] Finkelstein EA, Trogdon JG, Cohen JW, Dietz W. Annual medical spending attributable to obesity: payer-and service-specific estimates. Health Aff (Millwood). 2009 Sep-Oct;28(5):w822-31. doi: 10.1377/hlthaff.28.5.w822. Epub 2009 Jul 27. PMID 19635784
- [Background] Flegal KM. Epidemiologic aspects of overweight and obesity in the United States. Physiol Behav. 2005 Dec 15;86(5):599-602. doi: 10.1016/j.physbeh.2005.08.050. Epub 2005 Oct 19. PMID 16242735
- [Background] Flegal KM, Carroll MD, Ogden CL, Curtin LR. Prevalence and trends in obesity among US adults, 1999-2008. JAMA. 2010 Jan 20;303(3):235-41. doi: 10.1001/jama.2009.2014. Epub 2010 Jan 13. PMID 20071471
- [Background] Fontaine KR, Redden DT, Wang C, Westfall AO, Allison DB. Years of life lost due to obesity. JAMA. 2003 Jan 8;289(2):187-93. doi: 10.1001/jama.289.2.187. PMID 12517229
- [Background] Foster GD, Sherman S, Borradaile KE, Grundy KM, Vander Veur SS, Nachmani J, Karpyn A, Kumanyika S, Shults J. A policy-based school intervention to prevent overweight and obesity. Pediatrics. 2008 Apr;121(4):e794-802. doi: 10.1542/peds.2007-1365. PMID 18381508
- [Background] Green M, Scott N, Diyankova I, Gasser C. Eating disorder prevention: an experimental comparison of high level dissonance, low level dissonance, and no-treatment control. Eat Disord. 2005 Mar-Apr;13(2):157-69. doi: 10.1080/10640260590918955. PMID 16864339
- [Background] Green, H. J., Frank, R. M., Butwell, A., & Beck, O. J. (2007). Implementation and evaluation of brief cognitivebehavioural therapy in a mental health acute assessment and treatment service. Behaviour Change, 24(2), 87-98.
- [Background] Haines J, Neumark-Sztainer D, Wall M, Story M. Personal, behavioral, and environmental risk and protective factors for adolescent overweight. Obesity (Silver Spring). 2007 Nov;15(11):2748-60. doi: 10.1038/oby.2007.327. PMID 18070766
- [Background] Harris JK, French SA, Jeffery RW, McGovern PG, Wing RR. Dietary and physical activity correlates of long-term weight loss. Obes Res. 1994 Jul;2(4):307-13. doi: 10.1002/j.1550-8528.1994.tb00069.x. PMID 16358394
- [Background] Heil DP. Predicting activity energy expenditure using the Actical activity monitor. Res Q Exerc Sport. 2006 Mar;77(1):64-80. doi: 10.1080/02701367.2006.10599333. PMID 16646354
- [Background] Hill JO, Peters JC. Environmental contributions to the obesity epidemic. Science. 1998 May 29;280(5368):1371-4. doi: 10.1126/science.280.5368.1371. PMID 9603719
- [Background] Hoagwood K, Olin SS. The NIMH blueprint for change report: research priorities in child and adolescent mental health. J Am Acad Child Adolesc Psychiatry. 2002 Jul;41(7):760-7. doi: 10.1097/00004583-200207000-00006. PMID 12108799
- [Background] Hodgkins C, Frost-Pineda K, Gold MS. Weight gain during substance abuse treatment: the dual problem of addiction and overeating in an adolescent population. J Addict Dis. 2007;26 Suppl 1:41-50. doi: 10.1300/J069v26S01_05. PMID 19283973
- [Background] Jacobson NS, Truax P. Clinical significance: a statistical approach to defining meaningful change in psychotherapy research. J Consult Clin Psychol. 1991 Feb;59(1):12-9. doi: 10.1037//0022-006x.59.1.12. PMID 2002127
- [Background] Jiang J, Xia X, Greiner T, Wu G, Lian G, Rosenqvist U. The effects of a 3-year obesity intervention in schoolchildren in Beijing. Child Care Health Dev. 2007 Sep;33(5):641-6. doi: 10.1111/j.1365-2214.2007.00738.x. PMID 17725789
- [Background] Klohe DM, Clarke KK, George GC, Milani TJ, Hanss-Nuss H, Freeland-Graves J. Relative validity and reliability of a food frequency questionnaire for a triethnic population of 1-year-old to 3-year-old children from low-income families. J Am Diet Assoc. 2005 May;105(5):727-34. doi: 10.1016/j.jada.2005.02.008. PMID 15883549
- [Background] Lipsey, M. W., & Wilson, D. B. (2001). Practical meta-analysis. Thousand Oaks, CA: Sage
- [Background] Lowe MR, Annunziato RA, Markowitz JT, Didie E, Bellace DL, Riddell L, Maille C, McKinney S, Stice E. Multiple types of dieting prospectively predict weight gain during the freshman year of college. Appetite. 2006 Jul;47(1):83-90. doi: 10.1016/j.appet.2006.03.160. Epub 2006 May 2. PMID 16650913
- [Background] MacKinnon, D. P. (2008). Multivariate Applications: Introduction to Statistical Mediation Analysis. New York: Lawrence Erlbaum Associates.
- [Background] Martin M, Beekley A, Kjorstad R, Sebesta J. Socioeconomic disparities in eligibility and access to bariatric surgery: a national population-based analysis. Surg Obes Relat Dis. 2010 Jan-Feb;6(1):8-15. doi: 10.1016/j.soard.2009.07.003. Epub 2009 Jul 17. PMID 19782647
- [Background] Matusek JA, Wendt SJ, Wiseman CV. Dissonance thin-ideal and didactic healthy behavior eating disorder prevention programs: results from a controlled trial. Int J Eat Disord. 2004 Dec;36(4):376-88. doi: 10.1002/eat.20059. PMID 15558649
- [Background] McCarthy HD, Cole TJ, Fry T, Jebb SA, Prentice AM. Body fat reference curves for children. Int J Obes (Lond). 2006 Apr;30(4):598-602. doi: 10.1038/sj.ijo.0803232. PMID 16570089
- [Background] McMillan W, Stice E, Rohde P. High- and low-level dissonance-based eating disorder prevention programs with young women with body image concerns: an experimental trial. J Consult Clin Psychol. 2011 Feb;79(1):129-34. doi: 10.1037/a0022143. PMID 21261438
- [Background] Mitchell KS, Mazzeo SE, Rausch SM, Cooke KL. Innovative interventions for disordered eating: evaluating dissonance-based and yoga interventions. Int J Eat Disord. 2007 Mar;40(2):120-8. doi: 10.1002/eat.20282. PMID 17089413
- [Background] Muthén, L. K., & Muthén, B. O. (1998-2010). Mplus User's Guide (6th ed.). Los Angeles: Muthén & Muthén.
- [Background] Muthén, L. K., & Muthén, B. O. (2002). How to use a Monte Carlo study to decide on sample size and determine power. Structural Equation Modeling, 9, 599-620.
- [Background] Neumark-Sztainer D, Story M, Hannan PJ, Perry CL, Irving LM. Weight-related concerns and behaviors among overweight and nonoverweight adolescents: implications for preventing weight-related disorders. Arch Pediatr Adolesc Med. 2002 Feb;156(2):171-8. doi: 10.1001/archpedi.156.2.171. PMID 11814380
- [Background] Perez M, Becker CB, Ramirez A. Transportability of an empirically supported dissonance-based prevention program for eating disorders. Body Image. 2010 Jun;7(3):179-86. doi: 10.1016/j.bodyim.2010.02.006. Epub 2010 Mar 23. PMID 20335084
- [Background] Preacher KJ, Hayes AF. Asymptotic and resampling strategies for assessing and comparing indirect effects in multiple mediator models. Behav Res Methods. 2008 Aug;40(3):879-91. doi: 10.3758/brm.40.3.879. PMID 18697684
- [Background] Reilly JJ, Penpraze V, Hislop J, Davies G, Grant S, Paton JY. Objective measurement of physical activity and sedentary behaviour: review with new data. Arch Dis Child. 2008 Jul;93(7):614-9. doi: 10.1136/adc.2007.133272. Epub 2008 Feb 27. PMID 18305072
- [Background] Ricciardelli LA, McCabe MP. Dietary restraint and negative affect as mediators of body dissatisfaction and bulimic behavior in adolescent girls and boys. Behav Res Ther. 2001 Nov;39(11):1317-28. doi: 10.1016/s0005-7967(00)00097-8. PMID 11686266
- [Background] Richardson LP, Davis R, Poulton R, McCauley E, Moffitt TE, Caspi A, Connell F. A longitudinal evaluation of adolescent depression and adult obesity. Arch Pediatr Adolesc Med. 2003 Aug;157(8):739-45. doi: 10.1001/archpedi.157.8.739. PMID 12912778
- [Background] Roehrig M, Thompson JK, Brannick M, van den Berg P. Dissonance-based eating disorder prevention program: a preliminary dismantling investigation. Int J Eat Disord. 2006 Jan;39(1):1-10. doi: 10.1002/eat.20217. PMID 16254869
- [Background] Rolls, B., & Barnett, R. (2000). Volumetrics: Feel full on fewer calories. New York, NY: Harper Collins
- [Background] Rolls, B., & Barnett, R. (2000). Volumetrics: Feel full on fewer calories. New York, NY: Harper Collins.
- [Background] Roy-Byrne PP, Sherbourne CD, Craske MG, Stein MB, Katon W, Sullivan G, Means-Christensen A, Bystritsky A. Moving treatment research from clinical trials to the real world. Psychiatr Serv. 2003 Mar;54(3):327-32. doi: 10.1176/appi.ps.54.3.327. PMID 12610239
- [Background] Schoeller DA, Ravussin E, Schutz Y, Acheson KJ, Baertschi P, Jequier E. Energy expenditure by doubly labeled water: validation in humans and proposed calculation. Am J Physiol. 1986 May;250(5 Pt 2):R823-30. doi: 10.1152/ajpregu.1986.250.5.R823. PMID 3085521
- [Background] Schwitzer, A., & Choate, L., (2007). College student needs and counseling responses. Journal of College Counseling, 10, 3-5.
- [Background] Seeley JR, Stice E, Rohde P. Screening for depression prevention: identifying adolescent girls at high risk for future depression. J Abnorm Psychol. 2009 Feb;118(1):161-170. doi: 10.1037/a0014741. PMID 19222322
- [Background] Seidel A, Presnell K, Rosenfield D. Mediators in the dissonance eating disorder prevention program. Behav Res Ther. 2009 Aug;47(8):645-53. doi: 10.1016/j.brat.2009.04.007. Epub 2009 May 3. PMID 19457474
- [Background] Singer, J. D., & Willett, J. B. (2003). Applied Longitudinal Data Analysis: Modeling Change and Event Occurrence. New York: Oxford University Press.
- [Background] Sirard JR, Kubik MY, Fulkerson JA, Arcan C. Objectively measured physical activity in urban alternative high school students. Med Sci Sports Exerc. 2008 Dec;40(12):2088-95. doi: 10.1249/MSS.0b013e318182092b. PMID 18981940
- [Background] Steele CM, Southwick LL, Critchlow B. Dissonance and alcohol: drinking your troubles away. J Pers Soc Psychol. 1981 Nov;41(5):831-46. doi: 10.1037//0022-3514.41.5.831. PMID 7299630
- [Background] Stice E, Whitenton K. Risk factors for body dissatisfaction in adolescent girls: a longitudinal investigation. Dev Psychol. 2002 Sep;38(5):669-78. doi: 10.1037//0012-1649.38.5.669. PMID 12220046
- [Background] Stice E, Cooper JA, Schoeller DA, Tappe K, Lowe MR. Are dietary restraint scales valid measures of moderate- to long-term dietary restriction? Objective biological and behavioral data suggest not. Psychol Assess. 2007 Dec;19(4):449-58. doi: 10.1037/1040-3590.19.4.449. PMID 18085937
- [Background] Stice E, Fisher M, Lowe MR. Are dietary restraint scales valid measures of acute dietary restriction? Unobtrusive observational data suggest not. Psychol Assess. 2004 Mar;16(1):51-9. doi: 10.1037/1040-3590.16.1.51. PMID 15023092
- [Background] Stice E, Marti CN, Rohde P, Shaw H. Testing mediators hypothesized to account for the effects of a dissonance-based eating disorder prevention program over longer term follow-up. J Consult Clin Psychol. 2011 Jun;79(3):398-405. doi: 10.1037/a0023321. PMID 21500884
- [Background] Stice E, Marti CN, Shaw H, Jaconis M. An 8-year longitudinal study of the natural history of threshold, subthreshold, and partial eating disorders from a community sample of adolescents. J Abnorm Psychol. 2009 Aug;118(3):587-97. doi: 10.1037/a0016481. PMID 19685955
- [Background] Stice E, Marti CN, Spoor S, Presnell K, Shaw H. Dissonance and healthy weight eating disorder prevention programs: long-term effects from a randomized efficacy trial. J Consult Clin Psychol. 2008 Apr;76(2):329-40. doi: 10.1037/0022-006X.76.2.329. PMID 18377128
- [Background] Stice E, Mazotti L, Weibel D, Agras WS. Dissonance prevention program decreases thin-ideal internalization, body dissatisfaction, dieting, negative affect, and bulimic symptoms: A preliminary experiment. Int J Eat Disord. 2000 Mar;27(2):206-17. doi: 10.1002/(sici)1098-108x(200003)27:23.0.co;2-d. PMID 10657894
- [Background] Stice E, Presnell K, Shaw H, Rohde P. Psychological and behavioral risk factors for obesity onset in adolescent girls: a prospective study. J Consult Clin Psychol. 2005 Apr;73(2):195-202. doi: 10.1037/0022-006X.73.2.195. PMID 15796626
- [Background] Stice E, Rohde P, Gau J, Shaw H. An effectiveness trial of a dissonance-based eating disorder prevention program for high-risk adolescent girls. J Consult Clin Psychol. 2009 Oct;77(5):825-34. doi: 10.1037/a0016132. PMID 19803563
- [Background] Stice E, Rohde P, Seeley JR, Gau JM. Brief cognitive-behavioral depression prevention program for high-risk adolescents outperforms two alternative interventions: a randomized efficacy trial. J Consult Clin Psychol. 2008 Aug;76(4):595-606. doi: 10.1037/a0012645. PMID 18665688
- [Background] Stice E, Rohde P, Shaw H, Gau J. An effectiveness trial of a selected dissonance-based eating disorder prevention program for female high school students: Long-term effects. J Consult Clin Psychol. 2011 Aug;79(4):500-8. doi: 10.1037/a0024351. PMID 21707136
- [Background] Stice E, Rohde P, Shaw H, Marti CN. Efficacy trial of a selective prevention program targeting both eating disorder symptoms and unhealthy weight gain among female college students. J Consult Clin Psychol. 2012 Feb;80(1):164-170. doi: 10.1037/a0026484. Epub 2011 Nov 28. PMID 22122289
- [Background] Stice E, Shaw H, Marti CN. A meta-analytic review of obesity prevention programs for children and adolescents: the skinny on interventions that work. Psychol Bull. 2006 Sep;132(5):667-91. doi: 10.1037/0033-2909.132.5.667. PMID 16910747
- [Background] Stice E, Shaw H, Marti CN. A meta-analytic review of eating disorder prevention programs: encouraging findings. Annu Rev Clin Psychol. 2007;3:207-31. doi: 10.1146/annurev.clinpsy.3.022806.091447. PMID 17716054
- [Background] Stice E, Shaw H, Burton E, Wade E. Dissonance and healthy weight eating disorder prevention programs: a randomized efficacy trial. J Consult Clin Psychol. 2006 Apr;74(2):263-75. doi: 10.1037/0022-006X.74.2.263. PMID 16649871
- [Background] Subar AF, Thompson FE, Kipnis V, Midthune D, Hurwitz P, McNutt S, McIntosh A, Rosenfeld S. Comparative validation of the Block, Willett, and National Cancer Institute food frequency questionnaires : the Eating at America's Table Study. Am J Epidemiol. 2001 Dec 15;154(12):1089-99. doi: 10.1093/aje/154.12.1089. PMID 11744511
- [Background] Surrao J, Sawaya AL, Dallal GE, Tsay R, Roberts SB. Use of food quotients in human doubly labeled water studies: comparable results obtained with 4 widely used food intake methods. J Am Diet Assoc. 1998 Sep;98(9):1015-20. doi: 10.1016/S0002-8223(98)00232-6. PMID 9739802
- [Background] Trost SG, McIver KL, Pate RR. Conducting accelerometer-based activity assessments in field-based research. Med Sci Sports Exerc. 2005 Nov;37(11 Suppl):S531-43. doi: 10.1249/01.mss.0000185657.86065.98. PMID 16294116
- [Background] Trost SG, Pate RR, Freedson PS, Sallis JF, Taylor WC. Using objective physical activity measures with youth: how many days of monitoring are needed? Med Sci Sports Exerc. 2000 Feb;32(2):426-31. doi: 10.1097/00005768-200002000-00025. PMID 10694127
- [Background] Turk MW, Yang K, Hravnak M, Sereika SM, Ewing LJ, Burke LE. Randomized clinical trials of weight loss maintenance: a review. J Cardiovasc Nurs. 2009 Jan-Feb;24(1):58-80. doi: 10.1097/01.JCN.0000317471.58048.32. PMID 19114803
- [Background] van Strien, T., Frijters, J. E., Van Staveren, W. A., Defares, P. B., & Deurenberg, P. (1986). The predictive validity of the Dutch Restrained Eating Scale. Int J Eat Disord, 5, 747-755
- [Background] Ward DS, Evenson KR, Vaughn A, Rodgers AB, Troiano RP. Accelerometer use in physical activity: best practices and research recommendations. Med Sci Sports Exerc. 2005 Nov;37(11 Suppl):S582-8. doi: 10.1249/01.mss.0000185292.71933.91. PMID 16294121
- [Background] Weisz JR, Donenberg GR, Han SS, Kauneckis D. Child and adolescent psychotherapy outcomes in experiments versus clinics: why the disparity? J Abnorm Child Psychol. 1995 Feb;23(1):83-106. doi: 10.1007/BF01447046. PMID 7759676
- [Background] Weyers AM, Mazzetti SA, Love DM, Gomez AL, Kraemer WJ, Volek JS. Comparison of methods for assessing body composition changes during weight loss. Med Sci Sports Exerc. 2002 Mar;34(3):497-502. doi: 10.1097/00005768-200203000-00017. PMID 11880815
- [Background] Wichstrom L. Psychological and behavioral factors unpredictive of disordered eating: a prospective study of the general adolescent population in Norway. Int J Eat Disord. 2000 Jul;28(1):33-42. doi: 10.1002/(sici)1098-108x(200007)28:13.0.co;2-h. PMID 10800012
- [Background] Wong SL, Colley R, Connor Gorber S, Tremblay M. Actical accelerometer sedentary activity thresholds for adults. J Phys Act Health. 2011 May;8(4):587-91. doi: 10.1123/jpah.8.4.587. PMID 21597132
- [Background] Yancey AK, Ortega AN, Kumanyika SK. Effective recruitment and retention of minority research participants. Annu Rev Public Health. 2006;27:1-28. doi: 10.1146/annurev.publhealth.27.021405.102113. PMID 16533107
- [Derived] Call CC, D'Adamo L, Butryn ML, Stice E. Examining weight suppression as a predictor and moderator of intervention outcomes in an eating disorder and obesity prevention trial: A replication and extension study. Behav Res Ther. 2021 Jun;141:103850. doi: 10.1016/j.brat.2021.103850. Epub 2021 Mar 29. PMID 33839586
- [Derived] Stice E, Desjardins CD, Shaw H, Rohde P. Moderators of two dual eating disorder and obesity prevention programs. Behav Res Ther. 2019 Jul;118:77-86. doi: 10.1016/j.brat.2019.04.002. Epub 2019 Apr 12. PMID 31005674
- [Derived] Rohde P, Arigo D, Shaw H, Stice E. Relation of self-weighing to future weight gain and onset of disordered eating symptoms. J Consult Clin Psychol. 2018 Aug;86(8):677-687. doi: 10.1037/ccp0000325. PMID 30035584
- [Derived] Rohde P, Desjardins CD, Arigo D, Shaw H, Stice E. Mediators of two selective prevention interventions targeting both obesity and eating disorders. Behav Res Ther. 2018 Jul;106:8-17. doi: 10.1016/j.brat.2018.04.004. Epub 2018 Apr 24. PMID 29715529
- [Derived] Stice E, Rohde P, Shaw H, Gau JM. An experimental therapeutics test of whether adding dissonance-induction activities improves the effectiveness of a selective obesity and eating disorder prevention program. Int J Obes (Lond). 2018 Mar;42(3):462-468. doi: 10.1038/ijo.2017.251. Epub 2017 Oct 9. PMID 28990590
- [Derived] Arigo D, Rohde P, Shaw H, Stice E. Psychosocial Predictors of Physical Activity Change Among College Students in an Obesity Prevention Trial. J Phys Act Health. 2017 Jul;14(7):513-519. doi: 10.1123/jpah.2016-0515. Epub 2017 Mar 14. PMID 28290744